CLINICAL TRIAL: NCT02480933
Title: Silent Breast Cancer A Study of the Disease Prevalence Held by Imaging Guided Biopsies in Autopsy Specimens
Acronym: SISYPHUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Hospitalar Lisboa Ocidental (Other Government)
Collaborators: Instituto Nacional de Medicina Legal e Ciências Forenses, Delegação do Sul (Unknown)
Responsible Party: Principal Investigator, Zacharoula Sidiropoulou, Zacharoula Sidiropoulou MD, MSc, Principal Investigator, General Surgery Assistent, Centro Hospitalar Lisboa Ocidental
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CentroHLO
Record Dates: First submitted 2015-06-17; First posted 2015-06-25 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Female Breast Cancer; Male Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male | interventions — Biopsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- female cadavers (Experimental): female cadavers above 40 years without known breast cancer Bilateral mastectomy Biopsy
  Interventions: Procedure: Bilateral mastectomy; Other: Biopsy
- Male cadavers (Experimental): male cadavers above 40 years without known breast cancer Bilateral mastectomy Biopsy
  Interventions: Procedure: Bilateral mastectomy; Other: Biopsy

INTERVENTIONS:
Procedure: Bilateral mastectomy — Bilateral mastectomy and imaging study of cadaveric breasts
Other: Biopsy — Biopsy of BI-RADS 3 and superior lesions

SUMMARY:
The aim of this study is to define silent breast cancer prevalence in both sexes and will be held by biopsies performed in imaging suspicious areas of the breast (ecography and mammography) in cadavers without known breast cancer.

DETAILED DESCRIPTION:
Cadavers of both sexes are going to be submitted to bilateral mastectomy. The specimens are going to be examined by palpation, ecography and mammography and all areas with (Breast Imaging Reporting and Data System) BI-RADS classification >= 3 are going to be biopsied.

Biopsy specimens are going to be processed by the pathology department and cancers are going to be identified and classified by their molecular type.

The investigators intend to know which is the disease reservoir in various ages.

ELIGIBILITY:
Inclusion Criteria:

* Female and male cadavers above 40 years

Exclusion Criteria:

* Known breast cancer
* Breast tissue accidental damage

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Silent breast cancer prevalence | 2 years
  To define the existing disease that did not caused death in both sexes

SECONDARY OUTCOMES:
Silent breast cancer prevalent molecular profile | 2 years
  To identify those molecular subgroups of the disease that remain silent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol: https://doi.org/10.3892/mco.20 — http://www.spandidos-publications.com/mco — feasibility of the protocol paper